CLINICAL TRIAL: NCT01987531
Title: Hemodynamic Effect of Temporary Biventricular Pacing After Mitral and/or Tricuspid Valve Surgery in Patients With Preoperative Biventricular Dysfunction
Brief Title: Temporary Biventricular Pacing
Acronym: BIPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 816482
Record Dates: First submitted 2013-11-05; First posted 2013-11-19 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Right Ventricular (RV) Dysfunction
Keywords: after open cardiac chamber cardiac surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- left ventricular epicardial pacing lead (Experimental): Enrolled patients will have a temporary left ventricular epicardial pacing lead placed in addition to the standard right ventricular and right atrial temporary epicardial pacing leads after open cardiac chamber cardiac surgery.
  Interventions: Other: left ventricular epicardial pacing lead

INTERVENTIONS:
Other: left ventricular epicardial pacing lead

SUMMARY:
The hypothesis of this study is that temporary biventricular pacing will improve hemodynamic performance in patients with right ventricular dysfunction after open cardiac chamber cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* mitral or tricuspid valve surgery patients identified as having preoperative Right Ventricular dysfunction and Left Ventricular Ejection Fraction less than 45 percent

Exclusion Criteria:

* Patients with in-situ biventricular pacemakers
* Pregnant or lactating females

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Right ventricular function of the heart | 24 hours after cardiac surgery completion
  Right Ventricular function is evaluated through combined echocardiographic interventricular synchrony variables which include pulmonary artery catheter derived cardiac index, pulmonary artery (PA) pressure, central venous pressure (CVP), CVP versus PA diastolic pressure, and systolic blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: William Vernick, MD, Principal Investigator — University of Pennsylvania, Anesthesia
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States